CLINICAL TRIAL: NCT05403164
Title: The Role of Epithelial-mesenchymal Transition in Patients With Periodontitis (An Immunohistochemistry Study)
Brief Title: Epithelial Mesenchymal Transition and Periodontitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Saif Sehaam Saliem, Professor, University of Baghdad
Other Study IDs: 241621
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Periodontitis; Periodontal Diseases; Epithelial-Mesenchymal Transition; Transcription Factors; Epithelial Attachment; Gram-Negative Bacteria
MeSH Terms: conditions — Periodontitis; Periodontal Diseases | interventions — Gingivectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontitis: Patients with periodontitis which is defined by interdental clinical attachment loss (CAL) ≥ 2 non-adjacent teeth, or Buccal or Oral CAL ≥ 3 mm with probing pocket depth (PPD) > 3 mm is detectable at ≥2 teeth. All patients should be indicated for periodontal surgery.
  Interventions: Procedure: Modified Widman flap
- Healthy periodontium: Healthy periodontium is defined by absence of CAL, PPD ≤3 mm, bleeding on probing <10%, and no evidence of radiological bone loss. Gingival samples are collected from subjects referred for gingivectomy for esthetic reasons such as crown lengthening, gummy smile or prior to teeth extraction for orthodontic treatment.
  Interventions: Procedure: Gingivectomy

INTERVENTIONS:
Procedure: Modified Widman flap — 1. Administration of anaesthesia
  2. First incision (reversed bevel incision), scalpel is placed at 45 degree, 2mm apical to gingival margin in coronal-apical direction until touching the bone and moved continuously around the teeth without any vertical releasing incisions
  3. Partial mobilization of the mucoperiosteal flap (full thickness flaps both facially and orally) within the attached gingiva to the alveolar crest
  4. Second incision (sulcular incision)
  5. Third incision (horizontal incision), also interdentally to remove the delineated tissue and all granulation tissue which is used later for analysis.
  6. Root surface debridement
  7. Flap adaptation, complete coverage interdentally and suturing.
  Groups: Periodontitis
Procedure: Gingivectomy — 1. Administration of anaesthesia
  2. Marking the base of the sulcus with pocket marker tweezer.
  3. First incision (gingivectomy incision), scalpel blade placed 1mm apical to the bleeding points and the incision should be beveled 45 degrees coronally.
  4. Second incision (interdental) to free the tissue which is used for analysis later.
  5. Debriding the area and applying periodontal pack.
  Groups: Healthy periodontium

SUMMARY:
Periodontitis is a chronic inflammatory disease results is destruction of the attachment apparatus of the teeth and ultimately tooth loss.

Epithelial-mesenchymal transition (EMT) is a process comprises of series of events that influence a polarized epithelial cell to undergo molecular/morphological changes leading to acquisition of mesenchymal cell phenotype. This process is responsible for suppressing epithelial-phenotype and it is known to be triggered by chronic exposure to inflammatory cytokines, Gram-negative bacteria, hypoxia, smoking, and hyperglycemia.

Both periodontitis and EMT share common risk factors/promoters; however, the role of EMT in the pathogenesis of periodontitis is not fully elucidated yet. Potential induction of EMT within periodontal pockets may disrupt epithelial barrier thus facilitating invasion of pathogenic periodontal pathogens to deeper tissues resulting in further tissue breakdown and non-resolving periodontal lesion.

DETAILED DESCRIPTION:
Periodontitis is a highly prevalent inflammatory disease affecting the attachment apparatus of the teeth, leading to progressive destruction of periodontal ligament and resorption of alveolar bone which if not treated, at early stages, it will lead to tooth loss. It is characterised by presence of a wide diversity of pathogenic bacteria, specifically Gram-negative anaerobes, that possess range of virulence factors responsible for triggering intense inflammatory response. Although this response is protective in nature; however, it leads to undesirable collateral damage to the surrounding tissues that is further aggravated by the aberrant immune response of the host.

Epithelial-mesenchymal transition (EMT) is a process comprises of series of events that influence a polarized epithelial cell to undergo molecular/morphological changes leading to acquisition of mesenchymal cell phenotype. EMT is modulated by range of regulatory pathways; mainly, downstream of TGF-β signaling activity which is evident in many developmental and pathological situations in which EMT is reported, including embryogenesis, inflammation and tumor metastasis. The hallmark of TGFβ signaling is up-regulation of Snail, an E-cadherin repressor. Overexpression of Snail has been found in various fibrotic diseases, including liver fibrosis and renal fibrosis.

E-cadherin is a calcium-dependent homophilic cell adhesion molecule expressed on the cell surfaces of epithelium and is a critical structure for stratification of squamous epithelia. The significant reduction in E-cadherin expression observed in the gingival epithelium during pocket formation and is believed to contribute to the pathogenesis of periodontal disease.

Vimentin is a type III intermediate filament (IF) protein that is expressed in mesenchymal cells. IF, along with tubulin-based microtubules and actin-based microfilaments, comprises the cytoskeleton. All IF proteins are expressed in a highly developmentally-regulated fashion; vimentin is the major cytoskeletal component of mesenchymal cells. Because of this, vimentin is often used as a marker of mesenchymal-derived cells or cells undergoing EMT during both normal development and metastatic progression.

β-catenin is a dual function protein, involved in regulation and coordination of cell-cell adhesion and gene transcription. β-catenin also acts as a morphogen in later stages of embryonic development. Together with TGF-β, an important role of β-catenin is to induce a morphogenic change in epithelial cells. It induces them to abandon their tight adhesion and assume a more mobile and loosely associated mesenchymal phenotype.

Role of EMT on compromising epithelial barrier function of periodontal pocket lining is not fully elucidated yet. Reported risk factors of EMT including prolonged exposure to cytokines, Gram-negative bacteria, tobacco and hypoxia are also relevant to periodontitis. Potential induction of EMT within periodontal pockets may disrupt epithelial barrier thus facilitating invasion of pathogenic periodontal pathogens to deeper tissues resulting in further tissue breakdown and non-resolving periodontal lesion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with generalized periodontitis, unstable, no risk factor
* Selected site should be indicated for surgical treatment by modified Widman flap in posterior area and these sites must exhibit periodontal pockets ≥ 5mm or pockets ≥ 4mm with BOP
* Plaque index score < 10%
* Never smoker or former smoker
* Not currently using systemic or local antimicrobials (at least in the last three months)
* Not currently using a mouth rinse
* In good general health with no evidence of any systemic disease
* Willing to consent

Exclusion Criteria:

* Have history of systemic disease e.g., diabetes mellitus
* Periodontal treatment in the last 6 months
* Current participation in other clinical trials
* Pregnant women
* Current smoker
* Not willing to sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants involved in this study are recruited from the patient attending to the Department of Periodontics, College of Dentistry, University of Baghdad. Those patients were treated non-surgically by the residents in the department. Primary endpoint of is assessed three months after completion of non-surgical therapy. Patients with persistent pockets at posterior teeth indicated for modified Widman flap are included in the study. Prior to enrollment, aims and details of the study are clearly explained to the patients who then asked to sign the consent form. All procedures in this study followed Helsinki declaration and its later amendments for conducting human researches.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment loss (CAL) | Measured at baseline only before conducting periodontal surgery
  CAL is a linear distance (in mm) from cemento-enamel junction to the base of the sulcus/periodontal pocket measured by using a periodontal probe, recorded at six sites per tooth namely; mesio-facial, mid-facial, disto-facial, mesio-oral, mid-oral, disto-oral.
Probing pocket depth (PPD) | Measured at baseline only before conducting periodontal surgery
  PPD is the distance (in mm) from the gingival margin to the base of the sulcus/periodontal pocket measured by using a periodontal probe, recorded at six sites per tooth namely; mesio-facial, mid-facial, disto-facial, mesio-oral, mid-oral, disto-oral.

SECONDARY OUTCOMES:
Bleeding on probing (BOP) | Measured at baseline only before conducting periodontal surgery
  BOP is measured by inserting a periodontal probe to the bottom of the gingival sulcus/periodontal pocket and moved gently along the tooth (root) surface. If bleeding occurs within 30 seconds after probing, the site is given score (1), and a negative score (0) for the non-bleeding site. BOP is recorded at six sites per tooth namely; mesio-facial, mid-facial, disto-facial, mesio-oral, mid-oral, disto-oral.
Immunohistochemical expression of EMT-related markers | Measured at baseline
  Immunohistochemical expressions of four EMT-related markers (E-cadherin, Snail1, vimentin, β-catenin) in gingival samples collected from patients with periodontitis and healthy periodontium are measured.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, University of Baghdad, Baghdad, Iraq